CLINICAL TRIAL: NCT06629402
Title: A Randomized, Double-Blind, Placebo-Controlled Crossover Study of PF614 on Analgesic Response in the Cold Pressor Test in Healthy Male Subjects
Brief Title: Assessment of PF614 Effects on Experimental Pain in the Cold Pressure Test (PF614-201)
Acronym: CPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ensysce Biosciences (Industry)
Collaborators: Dr. Vince Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PF614-201
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Acute Pain
Keywords: Cold Pressor Test; CPT; Experimental Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Methodology: This will be a randomized, double-blind, placebo-controlled, 2-way crossover study to evaluate the onset of analgesia following administration of single oral doses of PF614 or placebo. The study will consist of 2 phases: Screening and Treatment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- PF614 50 mg (Experimental): Oral 50 mg
  Interventions: Drug: PF614
- PF614 100 mg (Experimental): Oral 100 mg
  Interventions: Drug: PF614
- Placebo (Placebo Comparator): Inactive medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF614 — Experimental oxycodone prodrug
  Other Names: Oxycodone prodrug
  Arms: PF614 100 mg; PF614 50 mg
Drug: Placebo — Inactive medication
  Other Names: Control
  Arms: Placebo

SUMMARY:
The primary objective of the study is to evaluate the onset of analgesia following administration of a single oral dose of PF614 (50 mg or 100 mg) or placebo in healthy male subjects in an experimental pain model (cold pressor test [CPT]).

DETAILED DESCRIPTION:
Researchers will compare drug PF614 to a placebo (a look-alike substance that contains no drug) to see if drug PF614 works to prevent moderate-to-severe experimental pain.

Study subjects will:

* On the Screening Day: Immerse their non-dominant hand in an ice cold water bath to assess their baseline pain threshold. Subjects will report when they first feel pain (onset) and how long they can keep their hand immersed in ice-cold water (maximum = 3 minutes).
* On Treatment Day 1: Repeat the initial CPT test for pain, then take drug PF614 or a placebo capsule (the study will be blinded so they won't know which treatment they received). After taking a single dose of study medication, they will be tested again for when they first feel pain (onset) and how long they can keep their hand immersed in ice-cold water (maximum = 3 minutes) at 10 time periods up to 6 hours after taking the study medications.
* Report adverse events, if any.
* On Treatment Day 2: After a minimum of 5 days after Treatment Day 1, subjects will repeat the procedures from Treatment Day 1. They will receive the opposite medication that they received on Treatment Day 1 (this is a cross-over design). They will be tested again for when they first feel pain (onset) and how long they can keep their hand immersed in ice-cold water (maximum = 3 minutes) at 10 time periods up to 6 hours after taking the study medications.
* Report adverse events, if any.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoking males, ages 18-55 years, inclusive, in good general health.
2. Body mass index (BMI) within the range of 18.0 to 34.0 kg/m2, inclusive, and a minimum weight of 50.0 kg.
3. Subjects must have completed at least 2 CPTs at Screening (minimum 30 minutes apart or when the dorsal surface hand skin temperature had returned to baseline temperature [±2°C]), with both tests resulting in latency time of greater than 20 seconds and less than 120 seconds.
4. Subjects must have had prior therapeutic experience with use of opioids for analgesia without showing signs of opioid-induced vomiting, dysphoria, or clinically significant sedation.
5. Subjects must have agreed to use a double-barrier contraceptive method (condom and spermicide, or condom along with female partner's contraceptive method [oral, injectable, implanted, transdermal, or intrauterine device (IUD) with or without hormones]), or at least one partner was confirmed to be surgically sterile, or subject must have agreed to remain abstinent from heterosexual intercourse at the time of Screening, during the study, and for 90 days following the last administration of study drug. Subjects must have agreed to not donate sperm during the study and for 90 days following the last administration of study drug.
6. Subjects must have been able to speak, read, and understand English sufficiently to allow completion of all study assessments.
7. Subjects must have been able to provide written informed consent.
8. Subjects must have been willing and able to follow study instructions and been likely to complete all study requirements.

Exclusion Criteria:

1. Lifetime history or presence of substance or alcohol use disorder, as defined by the Diagnostic and Statistical Manual of Mental Disorders - Fifth Edition, Text Revision (DSM-V-TR).
2. History or presence of clinically significant abnormality, as assessed by physical examination, medical history, electrocardiograms (ECGs), vital signs, or laboratory values, which, in the opinion of an investigator, would have jeopardized the safety of the subject or the validity of the study results. Retesting may have been permitted at the discretion of an investigator.
3. History or presence of acute respiratory depression, chronic pulmonary disease, cor pulmonale, delirium tremens, central nervous system (CNS) depression, or increased cerebrospinal or intracranial pressure.
4. History or presence of peripheral neuropathy or significant trauma or injury to non-dominant hand.
5. Documented history of, or currently active, seizure disorder (excluding febrile seizures in childhood), history of clinically significant head injury or syncope of unknown origin.
6. History or presence of obstructive sleep apnea.
7. History of gastrointestinal disturbance requiring frequent use of antacids.
8. History of or presence of trypsin deficiency.
9. History of allergy or hypersensitivity to oxycodone, any other opioid or naloxone.
10. Positive urine drug screen (UDS) or alcohol screen at Screening and at check-in to each treatment period (Day -1).
11. Positive for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or human immunodeficiency virus (HIV).
12. Positive result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at check-in to each treatment period (Day -1). If a subject presented with a positive result, the subject may have been rescheduled at the discretion of the investigator and in agreement with the sponsor.
13. Evidence of clinically significant hepatic or renal impairment including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5 × the upper limit of normal (ULN). Retesting may have been permitted at the discretion of an investigator at Screening and at admission to Treatment Period 1 (Day -1).
14. Use of prescription drugs and natural health products (e.g., herbal remedies) within at least 14 days or at least 5 times the t½ of the drug (if known), prior to first study drug administration in the Treatment Phase, whichever was longer.
15. Use of non-prescription (over-the-counter) drugs within at least 7 days or at least 5 times the t½ of the drug (if known), prior to first study drug administration in the Treatment Phase, whichever was longer. On a case-by-case basis, the medical monitor may have allowed some over-the-counter medications within the 7 day window if the t½ of the drug was short.
16. Use of any enzyme-modifying drugs or products, including strong inhibitors of cytochrome P450 (CYP) enzymes (e.g., clarithromycin, itraconazole, ketoconazole, nefazodone, posaconazole, telithromycin, voriconazole, cimetidine, fluoxetine, quinidine, erythromycin, ciprofloxacin, fluconazole, diltiazem and HIV antivirals) and strong inducers of CYP enzymes (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort) within 30 days of first study drug administration in the Treatment Phase.
17. Use of investigational drugs within at least 30 days or 5 times the t½ of the drug (if known), whichever was longer, prior to first study drug administration in the Treatment Phase.
18. Use of tobacco- or nicotine-containing products in the 3 months prior to Screening.
19. Donation or loss of blood in excess of 500 mL within 56 days prior to Screening, or plasma within 7 days prior to Screening.
20. Subject was an employee of the sponsor, a research site staff member directly affiliated with this study, or was an immediate family member, defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
21. Any other condition that, in an investigator's opinion, (i) put the subject at increased risk, (ii) could have confounded the study results, (iii) may have interfered significantly with the subject's participation in the study, or (iv) had the potential to limit the subject's ability to complete the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 16 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (pre-dose) in Time to Pain Onset (defined as time to first pain) | 6 hours
  The time to first pain was recorded by trained site staff using a stop watch. Each subject was instructed to remove their hand at 3 minutes if they had not yet reached pain tolerance. Separate assessments were made at pre-dose (within 60 minutes prior to dosing; at least duplicate measurements, 30 minutes apart) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, and 6 hours post-dose.
Change from Baseline in Pain Tolerance (defined as latency time required for removal of hand from water bath) | 6 hours
  The latency time to hand removal from the water bath was recorded by trained site staff using a separate stopwatch. Separate assessments were made at pre-dose (within 60 minutes prior to dosing; at least duplicate measurements, 30 minutes apart) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, and 6 hours post-dose.

SECONDARY OUTCOMES:
Change from Baseline in Maximum Pain Intensity (pain NRS) | 6 hours
  A pain intensity score (maximum pain intensity = most intense pain felt during the immersion period) was rated on an 11-point numerical rating scale (NRS) after the subject removed their hand. Each subject was instructed to remove their hand at 3 minutes if they had not yet reached pain tolerance. Separate assessments were made at pre-dose (within 60 minutes prior to dosing; at least duplicate measurements, 30 minutes apart) and at 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, and 6 hours post-dose.

OTHER OUTCOMES:
Change from Baseline in Dorsal Skin Temperature of the hand used in the CPT | 6 hours
  Dorsal surface temperature of hand used for CPT test was measured within 2 minutes of each CPT test.
Safety Endpoints | 3 days
  Treatment-Emergent Adverse Events
Safety Endpoints | 3 days
  Serious adverse events (SAEs)
Safety Endpoints | 3 days
  AEs leading to discontinuation
Safety Endpoints | 3 days
  Changes in systolic and diastolic blood pressure (mmHg)
Safety Endpoints | 3 days
  Changes in pulse rate (beats per minute)
Safety Endpoints | 3 days
  Changes in body temperature (ºC)
Safety Endpoints | 3 days
  Changes in respiratory rate (breaths per minute)
Safety Endpoints | 3 days
  Changes in oxygen saturation (SpO2)

CONTACTS AND LOCATIONS:
Overall Officials: William K Schmidt, PhD, Study Director — Ensysce Biosciences Inc.
Locations (1):
- Dr. Vince Clinical Research, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirkpatrick DL, Schmidt WK, Morales R, Cremin J, Seroogy J, Husfeld C, Jenkins T. In vitro and in vivo assessment of the abuse potential of PF614, a novel BIO-MD prodrug of oxycodone. J Opioid Manag. 2017 Jan/Feb;13(1):39-49. doi: 10.5055/jom.2017.0366. PMID 28345745
- [Background] Kirkpatrick DL, Evans C, Pestano LA, Millard J, Johnston M, Mick E, Schmidt WK. Clinical evaluation of PF614, a novel TAAP prodrug of oxycodone, versus OxyContin in a multi-ascending dose study with a bioequivalence arm in healthy volunteers. Clin Transl Sci. 2024 Mar;17(3):e13765. doi: 10.1111/cts.13765. PMID 38511523